CLINICAL TRIAL: NCT01573871
Title: Tolerance and Compliance of Infants Fed an Extensively Hydrolyzed Infant Formula
Brief Title: Tolerance and Compliance of Infants Fed an Hydrolyzed Infant Formula
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK94
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Infant; Gastrointestinal Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydrolyzed infant formula (Experimental): Hydrolyzed infant formula to be fed ad libitum
  Interventions: Other: Experimental Hydrolyzed infant formula

INTERVENTIONS:
Other: Experimental Hydrolyzed infant formula — Experimental hydrolyzed infant formula to be fed ad libitum

SUMMARY:
The objective of the study is to assess gastrointestinal tolerance and compliance in infants who require a hydrolyzed formula.

ELIGIBILITY:
Inclusion Criteria:

* Infant is 0 to 180 days of age
* Infant with persistent feeding intolerance symptoms; has had at least 1 formula switch OR infant is experiencing/being managed with an extensively hydrolyzed formula for suspected food protein intolerance or allergy or other condition where an extensively hydrolyzed formula is deemed appropriate
* Infant has not consumed an extensively hydrolyzed infant formula
* Use of prescription medications, OTC medications, home remedies, herbal preparations or rehydration fluids restricted
* Infant is not receiving steroids.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* Parent(s) confirm their intention not to administer solid foods or juices to their infant through the duration of the study.
* Parent(s) confirm their intention not to administer vitamin or mineral during the study

Exclusion Criteria:

• Participation in another study

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Weight maintenance | 14 days

SECONDARY OUTCOMES:
Formula volume intake | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, Study Chair — Abbott Nutrition
Locations (3):
- United States (3):
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Metro-Health Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, Huber Heights, Ohio